CLINICAL TRIAL: NCT00961909
Title: A Multi-Center, Randomized, Double-Blind, Multiple Ascending Dose, Placebo-Controlled, Parallel Group, 2-Part Study to Investigate the Safety, Tolerability, PK, and PD of Once Weekly RO5095932 in Patients With Type 2 Diabetes Mellitus on a Stable Dose of Metformin
Brief Title: A Study of RO5095932 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP22340
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1active (Experimental)
  Interventions: Drug: RO5095932; Drug: metformin
- 1placebo (Placebo Comparator)
  Interventions: Drug: metformin; Drug: placebo
- 2active (Experimental)
  Interventions: Drug: RO5095932; Drug: metformin
- 2placebo (Placebo Comparator)
  Interventions: Drug: metformin; Drug: placebo

INTERVENTIONS:
Drug: RO5095932 — cohorts receiving multiple ascending doses, sc once weekly for 4 weeks
  Arms: 1active
Drug: RO5095932 — dose titration to target dose, sc once weekly for 6 weeks
  Arms: 2active
Drug: metformin — stable dose
Drug: placebo — sc once weekly for 4 weeks
  Arms: 1placebo; 2placebo

SUMMARY:
This randomized, double-blind, placebo-controlled study will assess the efficacy, safety, tolerability, pharmacokinetics and pharmacodynamics of RO5095932 in patients with type 2 diabetes mellitus. Patients will be randomized to receive either RO5095932 subcutaneously once weekly or placebo for 4 weeks (part 1) or 6 weeks (part 2), in addition to their current stable doses of metformin.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-65 years of age
* females who are either surgically sterile or post-menopausal
* type 2 diabetes treated with a stable dose of metformin
* BMI between 25-39kg/m2
* HbA1c between 7 and 10%
* fasting plasma glucose between 7 and 13.3mmol/L

Exclusion Criteria:

* history of clinically significant cardiovascular disease
* history of clinically significant hepatic or renal disease or impairment
* recent therapy with insulin, thiazolidinedione, glucagon-like peptide-1 analogues, amylin analogues and/or DPP-IV inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: AEs, laboratory parameters, ECG, body weight, vital signs | monitored throughout study, with weekly ECG and 2x weekly to 2-weekly laboratory assessments on study treatment and at intervals during follow-up
Change in hemoglobin A1c (HbA1c) | from baseline to week 6

SECONDARY OUTCOMES:
Pharmacokinetics: blood concentration of RO5095932 after multiple dosing | multiple sampling weeks 1-4 or 1-6 respectively, and weekly during follow-up
Change in metabolic parameters: glucose, insulin, C-peptide | assessed after 4 or 6 weeks on study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (5):
  - Anaheim, California
  - Chula Vista, California
  - Fort Myers, Florida
  - Miramar, Florida
  - San Antonio, Texas